CLINICAL TRIAL: NCT06156449
Title: Effect of Thyme Oil on Respiratory Symptoms and Hemodynamic Parameters in COPD Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Zeliha CENGİZ, Associate Professor, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023/4947
Record Dates: First submitted 2023-11-15; First posted 2023-12-05 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Patient Engagement
Keywords: hemodynamic parameters; thyme oil; respiratory symptoms; COPD patients
MeSH Terms: conditions — Patient Participation; Signs and Symptoms, Respiratory | interventions — thyme oil

STUDY DESIGN:
Intervention Model Description: In the study, patients will be stratified according to their gender (male and female) status and the blocking process will be performed. In this study, block randomization will be done according to age groups in order to assign the participants to the experimental and control groups. Patients will be listed according to the hospitalization list and numbered up to 140. Numbers will be assigned to the experimental and control groups according to the random numbers list. Thus, the probability of each patient in the groups being in either of the intervention or control groups will be equalized.
  Group 1: experimental 2. Group: Control
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): No intervention will be applied to the control group and the measurements will be recorded simultaneously.
- experimental group (Experimental): After filling out the forms, thyme oil aromatherapy will be applied to the patients assigned to the experimental group .The oregano oil to be prepared must have a high carvacrol ratio. Thyme oil with a carvacrol ratio of at least 74% will be specific to each patient and will be given to the patient in the form of an inhaler stick. According to expert opinion; The patient's own room should be visited every 8 hours and the patient-specific inhaler stick should be sniffed into 8 breathing lungs. Each patient will use an inhaler stick for 5 days. Hemodynamic parameters (ph, CO 2, O 2 ) and COPD symptom will be measured before the intervention with the patient (pretest) and at the end of the 5th day (posttest). Vital signs will be measured and recorded three times a day in the patient's room at 08:00, 16:00 and 24:00.
  Interventions: Other: Thyme oil

INTERVENTIONS:
Other: Thyme oil — The composition of NV-2016 Coded Thyme Essential oil (Origanum vulgare) (GC-201900528) was obtained with Nature&Nurture (10 µL) macra (Barcode No: 8697742121135, Registration No: 381751). Content of origanum vulgare oil used: 1.3% y-Terpinene, 2.7% p-Cymene, 5.6% linalool, 1.2% terpinen-4-ol, 1.2 borneol, 1.2% β-Bisabolene Contains 3.2% tymol and 75.7% carvacrol.
  Arms: experimental group

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a high-prevalence, preventable and treatable disease characterized by abnormal respiratory symptoms and airway obstruction, often resulting from exposure to hazardous substances due to airway and/or alveolar abnormalities. The disease is an important problem with high morbidity and mortality rates all over the world and in our country. COPD is known as the third disease with a high mortality rate and the sixth disabling disease worldwide. The Global Burden of Disease Study reports 251 million cases of COPD worldwide in 2016. According to World Health Organization (WHO) data, it is estimated that 3.17 million deaths were caused by COPD in 2015. This number constitutes 5% of all deaths. More than 90% of these deaths occur in low- and middle-income countries.It has become common to use medicinal plants together with medical antiviral treatments to reduce the negative effects of COPD. Pulmonary elimination of thymol has been reported to have beneficial effects on respiratory diseases.

Our research is the first to investigate in detail the effects of thyme oil on the symptoms and hemodynamic parameters of COPD. The widespread use of the thyme plant among patients shows that the research is important because it is an easily accessible, cheap and reliable essential oil.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease is treated with pharmacological and non-pharmacological methods. The first step of disease management is pharmacological treatment. Pharmacological treatment is generally preferred to reduce the frequency, duration and severity of symptoms experienced by the patient, reduce the acute exacerbation of the disease, improve the exercise capacity of the patients and increase the quality of life. Non-pharmacological treatments are; These are practices such as physical therapy, massage, relaxation techniques, meditation, reiki, yoga, prayer, multivitamins, herbal medicines, osteopathy, cryopathy, homeopathy, acupuncture, acupressure, reflexology, music therapy, visualization, hypnosis, and suggestion.

It has become common to use medicinal plants together with medical antiviral treatments to reduce the negative effects of COPD. Among these, thyme is a plant from the Lamiaceae family that has no known significant side effects and is used for its healing effects. Thyme plant belongs to the mint family and the plant contains antioxidant compounds such as phenolic, eugenol, carvacrol and thymol. Pulmonary elimination of thymol has been reported to have beneficial effects on respiratory diseases. In the literature, Chabok et al. It has been reported that it improves gas exchange in the respiratory tract and increases oxygen saturation value. Similarly, Schönknecht et al. determined that thyme is a spasmolytic, antimicrobial, anti-inflammatory, immunomodulatory and antioxidant agent. Additionally, Oliveiro et al. reported that thyme could be an effective treatment of chronic diseases based on inflammatory processes in cases of morbidity and mortality in lung cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized with the diagnosis of COPD in the chest diseases service of a Training and Research Hospital located in the east of Turkey,
* Receiving the patient on the first day of admission to the chest diseases service (Day 1).
* Those who have been hospitalized in the chest diseases service for at least 3 days,
* Over 18 years of age,
* Being conscious,
* Open to communication and cooperation,
* Patients who volunteer to participate in the study will be included in the study.

Exclusion Criteria:

* Under 18 years of age,

  * Those with dementia and/or other organic mental disorders,
  * Those with mental retardation detected by clinical interview,
  * Those who have received any psychiatric diagnosis,
  * Those who are pregnant,
  * Those who do not want to participate in the research,
  * Patients transferred to intensive care or discharged will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-03-15 (Estimated); Study Completion 2024-04-15 (Estimated)

PRIMARY OUTCOMES:
Patient Introduction Form | 4 months
  This form, prepared by the researchers, consists of 13 questions about age, weight, gender, marital status, education status, employment status, income status, occupation and COPD characteristic.
COPD Symptom Form | 4 months
  This form, used by researchers with the support of the literature, consists of questions measuring the presence and severity of COPD symptoms.
The pH level | 4 months
  Hemodynamic Parameters
Level of O 2 | 4 months
  Hemodynamic Parameters
Level of CO 2 | 4 months
  Hemodynamic Parameters
Level of SaO 2 | 4 months
  Hemodynamic Parameters
pulse rate | 4 months
  Vital Signs Form
respiratory rate | 4 months
  Vital Signs Form

CONTACTS AND LOCATIONS:
Locations (1):
- Batman Training and Research Hospital, Batman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No